CLINICAL TRIAL: NCT05627739
Title: An Observational Study of Mycophenolate Mofetil Combined With Glucocorticoid in the Treatment of Relapse Vogt-Koyanagi-Harada Disease
Brief Title: A Study of Mycophenolate Mofetil Combined With Glucocorticoid Therapy in Relapse Vogt-Koyanagi-Harada Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Xiaomin Zhang, Principal Investigator, MD, PhD, Tianjin Medical University
Other Study IDs: 2022KY-28
Record Dates: First submitted 2022-11-11; First posted 2022-11-28 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Vogt-Koyanagi-Harada Disease; Mycophenolate Mofetil
MeSH Terms: conditions — Uveomeningoencephalitic Syndrome | interventions — Mycophenolic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mycophenolate Mofetil therapy Group: An initial dose of 0.5-1.0g bid MMF was orally administered every day, glucocorticoid was started at a dose of 0.5-0.8 mg/kg/day and no more than 60 mg/day.
  Interventions: Drug: Mycophenolate Mofetil
- traditional therapy group: Patients were treated with glucocorticoids alone or glucocorticoids combined with Cyclosporine.

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Glucocorticoid is started at a dose of 0.5-0.8 mg/kg/day, and 60 mg daily was the highest dose. Mycophenolate mofetilwas is started at a dose of 0.5-1.0g bid.
  Groups: Mycophenolate Mofetil therapy Group

SUMMARY:
This project is designed to test the hypothesis that Mycophenolate Mofetil is clinically useful for patients with relapse Vogt-Koyanagi-Harada disease

DETAILED DESCRIPTION:
Approval of the study was obtained from the hospital's ethical committee. The study design and methodology followed the tenets of Declaration of Helsinki. All patients were provided with written informed consent and received a thorough explanation of the use of Mycophenolate Mofetil, its potential risks and benefits. This is a monocenter, cohort, observational study evaluating patients with relapse VKH divided into two groups: Mycophenolate Mofetil therapy group and traditional therapy group.

For Mycophenolate Mofetil therapy group, an initial dose of 0.5-1.0g bid MMF was orally administered every day, glucocorticoid was started at a dose of 0.5-0.8 mg/kg/day and no more than 60 mg/day. For the traditional therapy group, patients were treated with glucocorticoids alone or glucocorticoids combined with Cyclosporine. Study participants will be followed for up to one year to determine efficacy and side effects.

According to best corrected visual acuity (BCVA), anterior chamber and vitreous inflammation, optical coherence tomography (OCT), change in corticosteroid dose during the study period and so on. The investigators evaluate the anti-inflammatory and immunosuppressive effects of MMF in treatment of relapse VKH.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 to 70 years of age.
2. Subjects who do not have previous, active or latent tuberculosis (TB).
3. Subject must start Vogt-Koyanagi-Harada disease more than two months, and develop at least one recurrence.

Exclusion Criteria:

1. Subject with confirmed or suspected infectious uveitis, including but not limited to infectious uveitis due to TB, cytomegalovirus (CMV), Human T-Lymphotropic Virus Type 1 (HTLV-1), Whipple's disease, Herpes Zoster virus (HZV), Lyme disease, toxoplasmosis and herpes simplex virus (HSV).
2. Subject with corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the trial.
3. Subject has previous exposure to anti-tumor necrosis factor (TNF) therapy or any biologic therapy (except intravitreal anti-vascular endothelial growth factor [VEGF] therapy) with a potential therapeutic impact on non-infectious uveitis.
4. Subject has received Ozurdex® (dexamethasone implant) within 6 months prior to the Baseline visit.
5. Subject has received intravitreal anti-VEGF therapy within 45 days of the Baseline visit for Lucentis® (ranibizumab) or Avastin® (bevacizumab) or within 60 days of the Baseline visit for anti-VEGF Trap (aflibercept).
6. Subject has received intravitreal methotrexate within 90 days prior to the Baseline visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VKH patients were recruited from the uveitis centre of Tianjin Medical University Eye Hospital
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change In LogMAR Best Corrected Visual Acuity (BCVA) From Baseline to Each Visit. | 24 weeks
  The participant's best corrected visual acuity was measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart. On the logMAR scale, 0 is equivalent to 20/20 visual acuity, the range of normal vision is considered to be from -0.2 - 0.1; higher values indicate visual impairment.
Recurrence rate | 24 weeks
  The recurrence rates in Mycophenolate mofetil treatment group and control group

SECONDARY OUTCOMES:
Change in Anterior Chamber (AC) Cell Grade From Baseline to Each Visit | 24 weeks
  Slit lamp examinations were conducted at each visit to assess AC cell count. The number of AC cells observed within a 1 mm × 1 mm slit beam was used to determine the grade according to the Standardization of Uveitis Nomenclature (SUN) criteria:
  Grade 0 = < 1 cell Grade 0.5+ = 1 - 5 cells Grade 1+ = 6 - 15 cells Grade 2+ = 16 - 25 cells Grade 3+ = 26 - 50 cells Grade 4+ = > 50 cells.
Prednisone exposure | 12 months
  Cumulative prednisone dose and/or mean prednisone dose

CONTACTS AND LOCATIONS:
Locations (1):
- xiaomin Zhang, Tianjin, Tianjin Municipality, China